CLINICAL TRIAL: NCT03929198
Title: Population-Based Lifestyle Intervention: Translation of the Pritikin Program to the Community- Pilot Study Protocol
Brief Title: Translation of Pritikin Program to the Community
Acronym: Prit-TN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Pritikin Longevity Center (Unknown); Wellmont Health System (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1204508
Record Dates: First submitted 2019-04-24; First posted 2019-04-26 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Metabolic Syndrome; Obesity; Weight Loss; Hypertension; Hypercholesterolemia; Hypertriglyceridemia
Keywords: metabolic syndrome; obesity
MeSH Terms: conditions — Metabolic Syndrome; Obesity; Weight Loss; Hypertension; Hypercholesterolemia; Hypertriglyceridemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group participated in a 6-week Pritikin diet, exercise program, and behavioral modification.
  Interventions: Other: Healthy Lifestyle
- Control (No Intervention): This group did not receive any intervention.

INTERVENTIONS:
Other: Healthy Lifestyle — 6 week Diet, Exercise training, Behavioral modification
  Arms: Intervention

SUMMARY:
The broad, long-term aims of this scope of work are to investigate the effects of the Pritikin Program to the general population. The study will test the effects on individuals from the community with dysfunctional lipids, blood pressure and glycemic control. To assess the effectiveness of the Pritikin Program in the community, the effects of Pritikin lifestyle intervention on overall health will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Dysfunctional lipids, blood pressure and glycemic control determined at a screening visit:

  * Triglycerides > 150 mg/dL OR HDL <50 in females, <40 mg/dL in males
  * Systolic blood pressure ≥130 mmHg OR diastolic blood pressure ≥80 mmHg (or on hypertension medication)
  * HbA1c ≥5.7% or higher
* No diagnosis or treatment for cancer in the past year
* No diagnosis of mild cognitive impairment or dementia in the past year
* Ability to perform daily exercise, including aerobic activity and resistance exercise
* Non-smoker in the past year

Exclusion Criteria:

* Positive exercise stress test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Body Weight | 6 weeks
Blood Pressure | 6 weeks
Cholesterol | 6 weeks
Triglycerides | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States